CLINICAL TRIAL: NCT05401084
Title: Impact of Low Carbohydrate and Low Gluten Diet on Acromegaly Progression, Symptoms, Complications, and Treatment Outcomes
Brief Title: Diet in the Management of Acromegaly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Artak Labadzhyan, Assistant professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001851
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate (Active Comparator): Counseling, education, and implementation of low carbohydrate diet.
  Interventions: Other: Diet
- Low gluten (Active Comparator): Counseling, education, and implementation of low gluten diet.
  Interventions: Other: Diet
- Standard (No Intervention): No change/intervention in diet. Continuation of standard diet.

INTERVENTIONS:
Other: Diet — Macronutrient diet changes.
  Arms: Carbohydrate; Low gluten

SUMMARY:
Impact of low carbohydrate and low gluten diet on acromegaly progression, symptoms, complications, and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly.

Exclusion Criteria:

* Diet restrictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in insulin-like growth factor 1 (IGF-1). | 8 weeks
  Change in IGF-1 will be assessed from baseline (pre-intervention) to end of follow up.
Change in growth hormone level (GH). | 8 weeks
  Change in GH level will be assessed from baseline (pre-intervention) to end of follow up.
Change in acromegaly related symptoms. | 8 weeks
  Change in acromegaly related symptoms will be assessed from baseline (pre-intervention) to end of follow up using Acromegaly Quality of Life Questionnaire (AcroQoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No